CLINICAL TRIAL: NCT03602638
Title: Chinese PLA General Hospital Hainan Branch
Brief Title: Effects of a Dipeptidyl Peptidase-4 Inhibitor Sitagliptininsulin on the Progression of Coronary Atherosclerosis in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Bo, Li Bo, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChinaPLAGH_hainan
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Atherosclerosis Type 2 Diabetes Mellitus Dipeptidyl Peptidase-4 Inhibitor GLP-1
MeSH Terms: interventions — Sitagliptin Phosphate; Acarbose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental)
  Interventions: Drug: Sitagliptin
- CONTROL (Active Comparator): Acarbose
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100mg QD
  Arms: Sitagliptin
Drug: Acarbose — Acarbose
  Arms: CONTROL

SUMMARY:
This study was to investigate the Effect of Sitagliptin, a dipeptidyl peptidase-4 inhibitor, on progression of coronary atherosclerosis in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This study was to investigate the Effect of Sitagliptin, a dipeptidyl peptidase-4 inhibitor, on progression of coronary atherosclerosis in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18, < 80 years old, with type 2 diabetes mellitus and coronary heart disease.

Exclusion Criteria:

* Allergy or hypersensitivity to any of the drug's components. Severe liver failure, moderate or severe kidney failure Malignant disease. Active infectious disease. Pregnancy or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
coronary calcification score | Changes from baseline in coronary calcification score at 18 months]
  Changes in coronary calcification score in Patients with coronary heart disease complicated with Type 2 Diabetes was measure with Computed tomography angiography. To measure the changes in coronary calcification score at 18 months.

IPD SHARING:
Plan to Share IPD: No